CLINICAL TRIAL: NCT01934803
Title: Zinc for HIV Disease Among Alcohol Users - an RCT in the Russia ARCH Cohort
Acronym: ZINC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jeffrey Samet, Chief, Section of General and Internal Medicine, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-31901; U01AA021989 (NIH)
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: HIV Infection; Alcohol Use
Keywords: Alcohol Use; Microbial Translocation; Inflammation; Altered Coagulation; Russia; Zinc; AMI; VACS index; Reynolds risk score
MeSH Terms: conditions — HIV Infections; Alcohol Drinking; Inflammation | interventions — gluconic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zinc gluconate (Active Comparator): Study participants will receive zinc gluconate supplements (15 mg for men and 12 mg for women) and will be instructed to take one pill daily for 18 months.
  Interventions: Dietary Supplement: Zinc gluconate
- Placebo (Placebo Comparator): Study participants will receive identically packaged placebo (sucrose) pills and will be instructed to take one pill daily for 18 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc gluconate — Study participants will be randomly assigned to a zinc gluconate or placebo group and will be instructed to take one pill of study medication orally daily for 18 months.
  Arms: Zinc gluconate
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This study is a double-blinded randomized controlled trial (RCT) to assess the efficacy of zinc supplementation vs. placebo among 250 HIV-infected Russians from the Russia ARCH Cohort, who are ART-naive at enrollment and have a recent history of heavy drinking.

DETAILED DESCRIPTION:
The combination of heavy alcohol consumption and HIV infection is associated with increased mortality, HIV disease progression, acute myocardial infarction (AMI) and a proinflammatory state characterized by increased biomarker levels of inflammation. Heavy alcohol use and HIV infection are both causes of microbial translocation, the process by which bacterial products from the gastrointestinal (GI) tract leak across the GI membrane to the portal circulation. Microbial translocation causes immune activation leading to end organ damage. Alcohol can cause microbial translocation via zinc deficiency. Zinc deficiency is common among HIV-infected heavy drinkers and linked to high mortality rates. Zinc supplementation is affordable, available, does not interfere with ART, and has minimal adverse drug reactions. In animal models zinc reduces ethanol associated microbial translocation. In human studies zinc slows HIV disease progression and reduces levels of inflammatory biomarkers which are strongly linked to mortality. Given zinc's potential efficacy we propose to conduct Zinc for INflammation and Chronic disease in HIV (ZINC HIV), a double-blinded randomized controlled trial to assess the efficacy of zinc supplementation vs. placebo among 250 HIV+ Russians, who are ART-naive at enrollment and have a recent history of heavy drinking. We will recruit most of our participants from the Russia cohort within the Uganda Russia Boston Alcohol Network for Alcohol Research Collaboration on HIV/AIDS (URBAN ARCH) Consortium study. Our specific aims will test the efficacy of zinc supplementation, compared to placebo to (1) improve markers of mortality as measured by the VACS index; (2) slow HIV disease progression as measured by CD4 cell count; (3) improve markers of AMI risk as measured by the Reynolds risk score; and (4) lower levels of microbial translocation and inflammation as measured by serum biomarkers. We hypothesize that as compared with placebo, patients receiving zinc supplementation will have significantly lower AMI and mortality risk as measured by the VACS index and Reynolds risk scores; higher CD4 cell counts; lower levels of biomarkers for microbial translocation and inflammation. Importantly, if our hypotheses are true, zinc supplementation could ultimately become a standard adjunctive therapy complementing alcohol interventions among HIV-infected persons even in resource limited environments. PUBLIC HEALTH RELEVANCE: The combination of heavy alcohol consumption and HIV infection results in serious health problems and an increased risk of death. Although it is not exactly clear how alcohol and HIV do this, inflammation appears to play an important role. Zinc supplementation has anti-inflammatory properties. This study is designed to see if giving zinc supplementation to HIV infected people who are heavy drinkers reduces the risk of serious health problems and death.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* HIV-infected
* ART naïve
* Heavy alcohol consumption [i.e., NIAAA at-risk drinking levels] in the past 30 days
* Provision of contact information for two contacts to assist with follow-up;
* Stable address within St. Petersburg or districts within 100 kilometers of St. Petersburg;
* Possession of a home or cellular telephone

Exclusion Criteria:

* Not fluent in Russian
* Cognitive impairment resulting in inability to provide informed consent based on assessor assessment
* Pregnancy
* Breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Improved markers of mortality as measured by change in VACS index | Participants will be followed for up to 18 months

SECONDARY OUTCOMES:
Slower HIV disease progression as measured by change in CD4 cell count | Participants will be followed for up to 18 months
Improved markers of AMI risk as measured by the Reynolds risk score | Participants will be followed for up to 18 months
Lower biomarker levels of microbial translocation and inflammation as measured by sCD-14, IL-6, D-dimer, IFABP, LBP | Participants will be followed for up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Samet, MD, MA, MPH, Principal Investigator — Boston Medical Center; Matthew S. Freiberg, MD, MSc, Principal Investigator — Vanderbilt University
Locations (1):
- Pavlov State Medical University, Saint Peterburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lodi S, Freiberg M, Gnatienko N, Blokhina E, Yaroslavtseva T, Krupitsky E, Murray E, Samet JH, Cheng DM. Per-protocol analysis of the ZINC trial for HIV disease among alcohol users. Trials. 2021 Mar 23;22(1):226. doi: 10.1186/s13063-021-05178-9. PMID 33757560
- [Derived] Freiberg MS, Cheng DM, Gnatienko N, Blokhina E, Coleman SM, Doyle MF, Yaroslavtseva T, Bridden C, So-Armah K, Tracy R, Bryant K, Lioznov D, Krupitsky E, Samet JH. Effect of Zinc Supplementation vs Placebo on Mortality Risk and HIV Disease Progression Among HIV-Positive Adults With Heavy Alcohol Use: A Randomized Clinical Trial. JAMA Netw Open. 2020 May 1;3(5):e204330. doi: 10.1001/jamanetworkopen.2020.4330. PMID 32383748
- [Derived] Gnatienko N, Freiberg MS, Blokhina E, Yaroslavtseva T, Bridden C, Cheng DM, Chaisson CE, Lioznov D, Bendiks S, Koerbel G, Coleman SM, Krupitsky E, Samet JH. Design of a randomized controlled trial of zinc supplementation to improve markers of mortality and HIV disease progression in HIV-positive drinkers in St. Petersburg, Russia. HIV Clin Trials. 2018 Jun;19(3):101-111. doi: 10.1080/15284336.2018.1459344. Epub 2018 Apr 17. PMID 29663871
- See also: Website for the Uganda, Russia, Boston Alcohol Network for Alcohol Research Collaboration on HIV/AIDS — http://www.urbanarch.org